CLINICAL TRIAL: NCT03828669
Title: Recovery Toolkits: An Observational Assessment of Nurse-Delivered, Pragmatic, Behavioral Pain Medicine for Post-Surgical Patients
Brief Title: Recovery Toolkits: Assessment of Pragmatic Behavioral Pain Medicine Delivered In Hospital After Surgery
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Beth Darnall, Principal Investigator, Stanford University
Other Study IDs: IDCP18RT
Record Dates: First submitted 2019-01-29; First posted 2019-02-04 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Post Surgical Pain
Keywords: behavioral medicine; pain; perioperative; enhanced recovery after surgery; surgery; intervention; post-operative pain; opioid; digital
MeSH Terms: conditions — Pain, Postoperative; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Usual Care: Prior to the roll-out of the Recovery Toolkit program, all post-surgical patients receiving current standard of care are given pain care surveys at hospital discharge. Survey questions ask about pain, and satisfaction with pain care. The investigators will conduct chart review for pain and opioid use.
- Recovery Toolkit: After launch of the Recovery Toolkit program on Jan 25, all post-surgical patients will be offered a Recovery Toolkit by a unit nurse. A pain survey will be administered at hospital discharge to assess about pain in the hospital, satisfaction with pain care, whether they received a Toolkit, use of the Toolkit, and likelihood to recommend the Toolkit. The investigators will conduct chart review for pain and opioid use.
  Interventions: Behavioral: Recovery Toolkits

INTERVENTIONS:
Behavioral: Recovery Toolkits — Recovery Toolkits are presented to patients in a branded bag and include a brochure, a self-help behavioral pain medicine book, a downloadable app, earbuds, and access to digital behavioral medicine (the "My Surgical Success" program including online educational videos)
  Groups: Recovery Toolkit

SUMMARY:
Behavioral pain medicine is largely absent from perioperative pathways, and on post-surgical recovery units. The goal of this project was to develop and implement "Recovery Toolkits", physical branded bags presented to patients after surgery. The "Recovery Toolkits" include a descriptive brochure and orientation to the contents of the bag. "Recovery Toolkits" include a behavioral pain medicine self-help book, an app with a downloadable pain management audiofile, earbuds, and a pen. Patients on each unit have access to iPads where they may view a digital behavioral pain medicine program ("My Surgical Success"), consisting of three 15-minute video learning modules. The "Recovery Toolkits" are psychologist-developed and nurse-delivered to every patient on the surgical recovery units. This pragmatic project seeks to understand:

1. Nurse perceived value of the intervention
2. Burden to nurses to deliver the intervention to all patients
3. Patient engagement with the Recovery Toolkits
4. Patient perceived value of the Recovery Toolkits
5. Patient satisfaction with pain care
6. Impact of Recovery Toolkits on pain and opioid use in hospital and at one-month discharge relative to a pre-Recovery Toolkit program cohort of patients.

DETAILED DESCRIPTION:
The Stanford "Recovery Toolkit" program is delivered by nurses across multiple surgical recovery units and surgery types, including neurosurgery, spine, and orthopedic surgeries. All patients who enter the units are offered a "Recovery Toolkit", which is a physical and branded bag. The program includes the following elements: a descriptive brochure and orientation to the contents of the bag. "Recovery Toolkits" include a behavioral pain medicine self-help book, an app with a downloadable pain management audiofile, earbuds, and a pen. Patients on all participating units have access to iPads where they may view a digital behavioral pain medicine program ("My Surgical Success"), consisting of three 15-minute video learning modules.

At discharge, patients are asked to evaluate their pain care and perception about the "Recovery Toolkit" in a 10-item survey that includes items as to whether the patient received a "Recovery Toolkit" (yes/no), did they use the "Recovery Toolkit" (yes/no), their satisfaction with the "Recovery Toolkit" (6-point likert scale), and recommendation for continuing the program (5-point likert scale). Chart review will extract data for demographics, surgery type, existing pain conditions and comorbidities, pain intensity scores averaged over the duration of their inpatient stay, as well as total opioid use during hospital stay and a daily average for inpatient opioid use. At one month after surgery, patients who agreed to be contacted will be asked their average pain intensity (0-10), whether they are taking opioid medication (yes/no) and how much (morphine equivalent daily dose), whether they have used the Recovery Toolkit information (yes/no), and, if yes, to please rate the helpfulness of the Recovery Toolkit information (0-10).

Nurses will be surveyed to determine the level of burden to deliver the intervention (0-6), their perceived value of the intervention to their patients (0-6), and their assessment on whether the program should be continued/expanded (0-6).

ELIGIBILITY:
Inclusion Criteria:

* Everyone

Exclusion Criteria:

* None, though Recovery Toolkits are English language

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Post-surgical inpatients (spine, neurosurgery, and other specialties)
Sampling Method: Non-Probability Sample
Enrollment: 649 (Actual)
Dates: Start 2019-01-25 (Actual); Primary Completion 2021-02-16 (Actual); Study Completion 2021-02-16 (Actual)

PRIMARY OUTCOMES:
Satisfaction with Recovery Toolkits | 10 minute survey administered at hospital discharge
  6-point scale
Likelihood to recommend | 10 minute survey administered at hospital discharge
  5-point scale

SECONDARY OUTCOMES:
Binary Opioid Use | Duration of inpatient hospital stay
  Average Morphine Equivalent Daily Dose
Average Pain | Duration of inpatient hospital stay
  Average of all pain ratings (0-10 numeric rating scale)
Opioid Daily Dose | 5 minuute survey administered 1 month after surgery
  Morphine Equivalent Daily Dose
Opioid use | 5 minute survey administered 1 month after surgery
  Binary question about continued opioid use (yes/no)
Average Pain Intensity | 5 minute survey administered 1 month after surgery
  Rating on 0-10 numeric rating scale
Opioid use | 5 minute survey administered 1 month after surgery
  Morphine Equivalent Daily Dose

CONTACTS AND LOCATIONS:
Overall Officials: Beth Darnall, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford Hospital, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No